CLINICAL TRIAL: NCT05879107
Title: A Phase III, Open-label, Randomized, Controlled, Multi-Country Study to Evaluate the Immune Response, Safety and Reactogenicity of RSVPreF3 OA Investigational Vaccine When Co Administered With PCV20 in Adults Aged 60\xa0Years and Older
Brief Title: Study to Assess the Immune Response, the Safety and the Reactogenicity of Respiratory Syncytial Virus (RSV) Prefusion Protein 3 Older Adult (OA) (RSVPreF3 OA) Investigational Vaccine When co Administered With PCV20 in Older Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 219276; 2022-501988-40-00 (Other: EU CTR number)
Record Dates: First submitted 2023-05-18; First posted 2023-05-30 (Actual); Results first posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: Respiratory syncytial virus; Vaccine; Older adult; Immunogenicity; Safety
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Co-administration Group (Experimental): Participants received both respiratory syncytial virus prefusion protein 3 older adult (RSVPreF3 OA) vaccine and 20-valent pneumococcal conjugate vaccine (PCV20) on Day 1.
  Interventions: Biological: RSVPreF3 OA investigational vaccine; Biological: PCV20
- Control Group (Active Comparator): Participants received PCV20 vaccine on Day 1 and RSVPreF3 OA vaccine on Day 31.
  Interventions: Biological: RSVPreF3 OA investigational vaccine; Biological: PCV20

INTERVENTIONS:
Biological: RSVPreF3 OA investigational vaccine — One dose of RSVPreF3 OA vaccine given intramuscularly in participant's non-dominant arm on Day 1 (in the Coad group) or Day 31(in the Control group).
  Other Names: RSVPreF3 OA
Biological: PCV20 — One dose of the 20-valent pneumococcal conjugate vaccine (PCV20) given intramuscularly in participant's dominant arm (Coad group) or non-dominant arm (Control group) on Day 1
  Other Names: 20 valent pneumococcal vaccine, Prevnar 20 (in US), Apexxnar (in Europe)

SUMMARY:
The purpose of this study is to assess the ability of RSVPreF3 OA investigational vaccine to generate an immune response when given in combination with PCV20 and its safety in older adults, aged ≥60 years of age.

ELIGIBILITY:
Inclusion Criteria:

* A male or female ≥60 years of age at the time of the first study intervention administration.
* Participants who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* Written or witnessed informed consent obtained from the participant prior to any study-specific procedure being performed.
* Participants living in the general community or in an assisted-living facility that provides minimal assistance, such that the participant is primarily responsible for self care and activities of daily living.
* Participants who are medically stable in the opinion of the investigator at the time of first study intervention administration. Participants with chronic stable medical conditions with or without specific treatment, are allowed to participate in this study if considered by the investigator as medically stable.

Exclusion Criteria:

* Any confirmed or suspected immunosuppressive or immunodeficient condition resulting from disease or immunosuppressive/cytotoxic therapy, based on medical history and physical examination.
* History of any reaction or hypersensitivity likely to be exacerbated by the study interventions, in particular any history of severe allergic reaction to any vaccine containing diphtheria toxoid, or pneumococcal polysaccharide 23-valent vaccine (PPSV23).
* Participants considered by investigator as suffering from serious or unstable chronic illness.
* Any history of dementia or any medical condition that moderately or severely impairs cognition.
* Recurrent or uncontrolled neurological disorders or seizures. Participants with medically controlled active or chronic neurological diseases can be enrolled in the study as per investigator assessment, provided that their condition will allow them to comply with the requirements of the protocol.
* Significant underlying illness that in the opinion of the investigator would be expected to prevent completion of the study.
* Any medical condition that in the judgment of the investigator would make intramuscular injection unsafe.
* History of previous vaccination with any licensed or investigational pneumococcal conjugate vaccine, or planned receipt through study participation.
* History of previous vaccination with any licensed or investigational pneumococcal polysaccharide vaccine in the last 5 years from enrollment, or planned receipt through study participation.
* Previous vaccination with any licensed or investigational RSV vaccine
* Use of any investigational or non-registered product (drug, vaccine or medical device) other than the study interventions during the period beginning 30 days before the first dose of study interventions and ending 30 days after the last study intervention administration, or their planned use during the study period.
* Planned or actual administration of a vaccine not foreseen by the study protocol in the period starting 30 days before the first study intervention administration and ending 30 days after the last study intervention administration. In the case of COVID 19 and inactivated/subunit influenza vaccines, this time window can be decreased to 14 days before and after each study intervention administration. In case of COVID-19 vaccine administration within 14 to 30 days window, the administration of COVID-19 vaccine should be in accordance with local government recommendations.

  * Planned or actual administration of adjuvanted quadrivalent influenza vaccine or live influenza vaccine not foreseen by the study protocol in the period starting 30 days before the first study intervention administration and ending 30 days after the last study intervention administration.

Note: In case an emergency mass vaccination for an unforeseen public health threat (e.g., a pandemic) is recommended and/or organized by the public health authorities outside the routine immunization program, the time period described above can be reduced if necessary for that vaccine, provided it is used according to the local governmental recommendations and that the Sponsor or designee is notified accordingly.

* Administration of long-acting immune-modifying drugs or planned administration at any time during the study period.
* Administration of immunoglobulins and/or any blood products or plasma derivatives during the period starting 90 days before the administration of first dose of study interventions or planned administration during the study period.
* Chronic administration (defined as more than 14 consecutive days in total) of immunosuppressants or other immune-modifying drugs during the period starting 90 days prior to the first study intervention dose or planned administration during the study period. For corticosteroids, this will mean prednisone ≥20 mg/day, or equivalent. Inhaled and topical steroids are allowed.
* Concurrently participating in another clinical study, at any time during the study period, in which the participant has been or will be exposed to an investigational or a non-investigational vaccine/product (drug or invasive medical device).
* History of chronic alcohol consumption and/or drug abuse as deemed by the investigator to render the potential participant unable/unlikely to provide accurate safety reports or comply with study procedures.
* Bedridden participants.
* Planned move during the study conduct that prohibits participation until EoS.
* Participation of any study personnel or their immediate dependents, family, or household members.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1113 (Actual)
Dates: Start 2023-05-26 (Actual); Primary Completion 2023-12-06 (Actual); Study Completion 2024-05-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (35):
- United States (20):
  - GSK Investigational Site, Guntersville, Alabama
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Modesto, California
  - GSK Investigational Site, Hamden, Connecticut
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, DeLand, Florida
  - GSK Investigational Site, Jupiter, Florida
  - GSK Investigational Site, Largo, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, West Des Moines, Iowa
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, Troy, Michigan
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, North Charleston, South Carolina
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Frisco, Texas
  - GSK Investigational Site, Mesquite, Texas
  - GSK Investigational Site, Plano, Texas
- Belgium (6):
  - GSK Investigational Site, Antwerp
  - GSK Investigational Site, Ghent
  - GSK Investigational Site, Kluisbergen
  - GSK Investigational Site, Mechelen
  - GSK Investigational Site, Namur
  - GSK Investigational Site, Wetteren
- Poland (7):
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Lublin
  - GSK Investigational Site, Pu?awy
  - GSK Investigational Site, Staszów
  - GSK Investigational Site, Warsaw
  - GSK Investigational Site, Wroclaw
- Spain (2):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Valencia

IPD SHARING:
Plan to Share IPD: Yes
GSK will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer tohttps://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in adult participants aged 60 years and older, in 38 study sites.
Pre-assignment Details: Out of 1113 participants, a total of 1110 were eligible and were randomized in a 1:1 ratio to either co-administration group or control group at Day 1.
Period: Overall Study
Arm/Group | Co-administration Group | Control Group
Started | 553 | 557
Completed | 539 | 531
Not Completed | 14 | 26
Not completed — Withdrawal by participant, not due to an adverse event | 5 | 7
Not completed — Migrated / moved from the study area | 1 | 1
Not completed — Lost to Follow-up | 8 | 13
Not completed — Death | 0 | 2
Not completed — Other | 0 | 3

BASELINE CHARACTERISTICS:
Population: Exposed set included all participants in the Enrolled set who received at least 1 study intervention.
Groups:
- Co-administration Group: Participants received both RSVPreF3 OA vaccine and PCV20 on Day 1.
- Total: Total of all reporting groups
Arm/Group | Co-administration Group | Control Group | Total
Number analyzed (Participants) | 553 | 557 | 1110
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.6 (7.28) | 69.6 (7.41) | 69.6 (7.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 316 | 315 | 631
  Male | 237 | 242 | 479
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — The "All Other Races" category (i.e., American Indian or Alaska Native and Asian) where 0<n<11 are combined into 1 category to maintain participant confidentiality and privacy.
  Participants
    Black or African American | 64 | 54 | 118
    All Other Races | 7 | 7 | 14
    White | 476 | 488 | 964
    Multiple | 2 | 4 | 6
    Other | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Geometric Mean Titers (GMT) of Opsonophagocytic (OP) Titers at 1 Month After the PCV20 Vaccination
Description: The OP titers were measured with multiplexed opsonophagocytosis assay and the results were expressed as GMT for each of the pneumococcal vaccine serotype.
Time Frame: At Day 31
Population: Per protocol set (PPS) for PCV20 included all eligible participants in the exposed set who: received the PVC20 vaccine, had immunogenicity results for OP titers, complied with blood draw interval, without intercurrent medical conditions and without prohibited concomitant medication/vaccination and who did not meet any of the criteria for elimination up to blood sample collection. Only participants with data available at the specified timepoint were included in the analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Co-administration Group | Control Group
Number analyzed (Participants) | 514 | 497
Titers
  Strep pneumoniae - serotype 1: number analyzed (Participants) | 513 | 497
  Strep pneumoniae - serotype 1 | 74.7 [64.1 to 87.1] | 110.8 [94.8 to 129.5]
  Strep pneumoniae - serotype 3 | 88.5 [78.3 to 99.9] | 116.2 [102.7 to 131.5]
  Strep pneumoniae - serotype 4: number analyzed (Participants) | 506 | 491
  Strep pneumoniae - serotype 4 | 1220.9 [1072.9 to 1389.3] | 1634.1 [1433.4 to 1862.8]
  Strep pneumoniae - serotype 5: number analyzed (Participants) | 512 | 497
  Strep pneumoniae - serotype 5 | 191.0 [159.9 to 228.1] | 260.3 [217.3 to 311.8]
  Strep pneumoniae - serotype 6A: number analyzed (Participants) | 512 | 493
  Strep pneumoniae - serotype 6A | 1790.0 [1527.8 to 2097.2] | 2458.3 [2091.8 to 2889.1]
  Strep pneumoniae - serotype 6B: number analyzed (Participants) | 509 | 492
  Strep pneumoniae - serotype 6B | 2121.6 [1839.0 to 2447.6] | 2996.9 [2590.3 to 3467.2]
  Strep pneumoniae - serotype 7F: number analyzed (Participants) | 511 | 496
  Strep pneumoniae - serotype 7F | 2411.3 [2154.1 to 2699.2] | 3225.1 [2876.2 to 3616.4]
  Strep pneumoniae - serotype 8: number analyzed (Participants) | 513 | 496
  Strep pneumoniae - serotype 8 | 522.9 [458.5 to 596.4] | 723.0 [632.5 to 826.5]
  Strep pneumoniae - serotype 9V: number analyzed (Participants) | 512 | 494
  Strep pneumoniae - serotype 9V | 937.0 [822.3 to 1067.8] | 1161.0 [1016.7 to 1325.8]
  Strep pneumoniae - serotype 10A: number analyzed (Participants) | 513 | 493
  Strep pneumoniae - serotype 10A | 6033.4 [5299.5 to 6868.9] | 7349.4 [6437.8 to 8389.9]
  Strep pneumoniae - serotype 11A: number analyzed (Participants) | 506 | 493
  Strep pneumoniae - serotype 11A | 798.0 [691.5 to 921.0] | 944.2 [816.9 to 1091.5]
  Strep pneumoniae - serotype 12F: number analyzed (Participants) | 507 | 487
  Strep pneumoniae - serotype 12F | 1608.4 [1382.9 to 1870.8] | 1932.4 [1656.5 to 2254.3]
  Strep pneumoniae - serotype 14: number analyzed (Participants) | 513 | 495
  Strep pneumoniae - serotype 14 | 2322.3 [2050.5 to 2630.1] | 3301.4 [2909.1 to 3746.7]
  Strep pneumoniae - serotype 15B: number analyzed (Participants) | 511 | 493
  Strep pneumoniae - serotype 15B | 4336.4 [3765.8 to 4993.5] | 6350.2 [5500.4 to 7331.3]
  Strep pneumoniae - serotype 18C | 1148.6 [997.6 to 1322.5] | 1480.0 [1282.4 to 1708.0]
  Strep pneumoniae - serotype 19A: number analyzed (Participants) | 513 | 495
  Strep pneumoniae - serotype 19A | 1392.3 [1244.3 to 1557.8] | 1933.8 [1725.2 to 2167.7]
  Strep pneumoniae - serotype 19F: number analyzed (Participants) | 509 | 494
  Strep pneumoniae - serotype 19F | 525.6 [461.6 to 598.5] | 696.7 [610.6 to 794.9]
  Strep pneumoniae - serotype 22F: number analyzed (Participants) | 510 | 495
  Strep pneumoniae - serotype 22F | 5492.3 [4788.1 to 6300.1] | 7351.5 [6397.0 to 8448.5]
  Strep pneumoniae - serotype 23F: number analyzed (Participants) | 514 | 495
  Strep pneumoniae - serotype 23F | 729.7 [613.0 to 868.6] | 995.0 [832.8 to 1188.7]
  Strep pneumoniae - serotype 33F | 14902.8 [13220.7 to 16798.8] | 20920.9 [18526.9 to 23624.3]
Statistical Analysis 1: Comparison: Co-administration Group vs Control Group; Strep pneumoniae - serotype 1; Test type: Non-Inferiority — NI was to be demonstrated if the upper limit of the 2-sided 95% confidence interval (CI) of the GMT ratio (as measured by the OP assay) between the Control group (at Day 31) versus Co-administration group (at Day 31) was <=2; GMT ratio = 1.48, 95% CI 2-sided [1.22 to 1.81] — The analysis of covariance (ANCOVA) model, for logarithm-transformed titers, included the treatment group and age category at vaccination as fixed effects and the pre-dose log-10 titer as covariate
Statistical Analysis 2: Comparison: Co-administration Group vs Control Group; Strep pneumoniae - serotype 3; Test type: Non-Inferiority — NI was to be demonstrated if the upper limit of the 2-sided 95% CI of the GMT ratio (as measured by the OP assay) between the Control group (at Day 31) versus Co-administration group (at Day 31) was <=2; GMT ratio = 1.31, 95% CI 2-sided [1.12 to 1.54] — The ANCOVA model, for logarithm-transformed titers, included the treatment group and age category at vaccination as fixed effects and the pre-dose log-10 titer as covariate
Statistical Analysis 3: Comparison: Co-administration Group vs Control Group; Strep pneumoniae - serotype 4; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; GMT ratio = 1.34, 95% CI 2-sided [1.13 to 1.58] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: Co-administration Group vs Control Group; Strep pneumoniae - serotype 5; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; GMT ratio = 1.36, 95% CI 2-sided [1.08 to 1.71] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Co-administration Group vs Control Group; Strep pneumoniae - serotype 6A; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; GMT ratio = 1.37, 95% CI 2-sided [1.12 to 1.69] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 6: Comparison: Co-administration Group vs Control Group; Strep pneumoniae - serotype 6B; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; GMT ratio = 1.41, 95% CI 2-sided [1.17 to 1.70] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 7: Comparison: Co-administration Group vs Control Group; Strep pneumoniae - serotype 7F; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; GMT ratio = 1.34, 95% CI 2-sided [1.16 to 1.55] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 8: Comparison: Co-administration Group vs Control Group; Strep pneumoniae - serotype 8; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; GMT ratio = 1.38, 95% CI 2-sided [1.17 to 1.64] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 9: Comparison: Co-administration Group vs Control Group; Strep pneumoniae - serotype 9V; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; GMT ratio = 1.24, 95% CI 2-sided [1.05 to 1.47] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 10: Comparison: Co-administration Group vs Control Group; Strep pneumoniae - serotype 10A; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; GMT ratio = 1.22, 95% CI 2-sided [1.03 to 1.44] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 11: Comparison: Co-administration Group vs Control Group; Strep pneumoniae - serotype 11A; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; GMT ratio = 1.18, 95% CI 2-sided [0.98 to 1.42] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 12: Comparison: Co-administration Group vs Control Group; Strep pneumoniae - serotype 12F; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; GMT ratio = 1.20, 95% CI 2-sided [0.99 to 1.46] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 13: Comparison: Co-administration Group vs Control Group; Strep pneumoniae - serotype 14; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; GMT ratio = 1.42, 95% CI 2-sided [1.21 to 1.67] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 14: Comparison: Co-administration Group vs Control Group; Strep pneumoniae - serotype 15B; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; GMT ratio = 1.46, 95% CI 2-sided [1.22 to 1.76] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 15: Comparison: Co-administration Group vs Control Group; Strep pneumoniae - serotype 18C; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; GMT ratio = 1.29, 95% CI 2-sided [1.07 to 1.55] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 16: Comparison: Co-administration Group vs Control Group; Strep pneumoniae - serotype 19A; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; GMT ratio = 1.39, 95% CI 2-sided [1.20 to 1.61] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 17: Comparison: Co-administration Group vs Control Group; Strep pneumoniae - serotype 19F; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; GMT ratio = 1.33, 95% CI 2-sided [1.12 to 1.57] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 18: Comparison: Co-administration Group vs Control Group; Strep pneumoniae - serotype 22F; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; GMT ratio = 1.34, 95% CI 2-sided [1.12 to 1.60] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 19: Comparison: Co-administration Group vs Control Group; Strep pneumoniae - serotype 23F; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; GMT ratio = 1.36, 95% CI 2-sided [1.09 to 1.71] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 20: Comparison: Co-administration Group vs Control Group; Strep pneumoniae - serotype 33F; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 2]; GMT ratio = 1.40, 95% CI 2-sided [1.20 to 1.64] — [estimate comment as in outcome 1, analysis 2]

2. Primary Outcome: Adjusted GMTs of Respiratory Syncytial Virus-A (RSV-A) Neutralizing Titers [Estimated Dilution 60 (ED60)] at 1 Month After the RSVPreF3 OA Vaccination
Description: Neutralizing titers were measured with neutralization assay and the results were expressed in ED60.
Time Frame: At Day 31 for Co-administration Group and at Day 61 for Control Group
Population: PPS for RSVPreF3 OA included all eligible participants in the exposed set who: received the RSVPreF3 OA vaccine, had immunogenicity results for RSV neutralizing titers, complied with blood draw interval, without intercurrent medical conditions and without prohibited concomitant medication/vaccination and who did not meet any of the criteria for elimination up to blood sample collection. Only the participants with RSV-A data at the specified timepoints were included in the analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Co-administration Group | Control Group
Number analyzed (Participants) | 512 | 382
Titers | 8338.2 [7639.0 to 9101.4] | 8872.7 [8038.2 to 9793.9]
Statistical Analysis 1: Comparison: Co-administration Group vs Control Group; RSV-A; Test type: Non-Inferiority — NI was to be demonstrated if the upper limit of the 2-sided 95% CI of the GMT ratio between the Control group (at Day 61) versus Co-administration group (at Day 31) for RSV-A neutralizing titer was <=1.5; GMT ratio = 1.06, 95% CI 2-sided [0.94 to 1.20] — [estimate comment as in outcome 1, analysis 2]

3. Primary Outcome: Adjusted GMTs of RSV-B Neutralizing Titers (ED60) at 1 Month After the RSVPreF3 OA Vaccination
Description: Neutralizing titers were measured with neutralization assay and the results were expressed in ED60.
Time Frame: At Day 31 for Co-administration Group and at Day 61 for Control Group
Population: PPS for RSVPreF3 OA. Only the participants with RSV-B data at the specified timepoints were included in the analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Co-administration Group | Control Group
Number analyzed (Participants) | 511 | 382
Titers | 9477.5 [8695.4 to 10329.9] | 9497.6 [8620.5 to 10463.9]
Statistical Analysis 1: Comparison: Co-administration Group vs Control Group; RSV-B; Test type: Non-Inferiority — NI was to be demonstrated if the upper limit of the 2-sided 95% CI of the GMT ratio between the Control group (at Day 61) versus Co-administration group (at Day 31) for RSV-B neutralizing titer was <=1.5; GMT ratio = 1.00, 95% CI 2-sided [0.89 to 1.13] — [estimate comment as in outcome 1, analysis 2]

4. Secondary Outcome: Mean Geometric Increase (MGI) of RSV-A Neutralizing Titers at 1 Month After the RSVPreF3 OA Vaccination
Description: The MGI was defined as the geometric mean increase of the within participant ratios of the post-vaccination titer over the pre-vaccination titer. Neutralizing titers were measured with neutralization assay.
Time Frame: At 1 month after the RSVPreF3 OA vaccine dose (Day 31 for Co-administration Group and Day 61 for Control Group) compared to Pre-vaccination (Day 1 for Co-administration Group and Day 31 for Control Group)
Population: PPS for RSVPreF3 OA. Only the participants with RSV-A data at the specified timepoints were included in the analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Co-administration Group | Control Group
Number analyzed (Participants) | 512 | 382
Ratio | 8.3 [7.6 to 9.1] | 9.3 [8.3 to 10.3]

5. Secondary Outcome: MGI of RSV-B Neutralizing Titers at 1 Month After the RSVPreF3 OA Vaccination
Description: as for outcome 4
Time Frame: as for outcome 4
Population: PPS for RSVPreF3 OA. Only the participants with RSV-B data at the specified timepoints were included in the analysis.
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Co-administration Group | Control Group
Number analyzed (Participants) | 511 | 382
Ratio | 9.4 [8.6 to 10.2] | 9.1 [8.2 to 10.1]

6. Secondary Outcome: Number of Participants With Solicited Administration Site Adverse Events (AEs) After Each Vaccine Dose Administration
Description: The solicited administration site events after vaccination include pain, erythema/redness, and swelling.
Time Frame: Within 7 days (the day of vaccination and 6 subsequent days) after each vaccine administration (vaccines administered at Day 1 for Co-Administration Group and at Days 1 and 31 for Control group)
Population: Exposed set included all participants in the Enrolled set who received at least 1 study intervention. Only those participants with solicited administration site AEs were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Co-administration Group | Control Group
Number analyzed (Participants) | 537 | 546
Participants
  Pain at injection site, PCV20 dose, given at Day 1 | 283 | 208
  Pain at injection site, RSV dose, given at Day 1: number analyzed (Participants) | 537 | 0
  Pain at injection site, RSV dose, given at Day 1 | 290 |
  Pain at injection site, RSV dose, given at Day 31: number analyzed (Participants) | 0 | 510
  Pain at injection site, RSV dose, given at Day 31 |  | 225
  Erythema at injection site, PCV20 dose, given at Day 1 | 24 | 21
  Erythema at injection site, RSV dose, given at Day 1: number analyzed (Participants) | 537 | 0
  Erythema at injection site, RSV dose, given at Day 1 | 54 |
  Erythema at injection site, RSV dose, given at Day 31: number analyzed (Participants) | 0 | 510
  Erythema at injection site, RSV dose, given at Day 31 |  | 33
  Swelling at injection site, PCV20 dose, given at Day 1 | 17 | 17
  Swelling at injection site, RSV dose, given at Day 1: number analyzed (Participants) | 537 | 0
  Swelling at injection site, RSV dose, given at Day 1 | 26 |
  Swelling at injection site, RSV dose, given at Day 31: number analyzed (Participants) | 0 | 510
  Swelling at injection site, RSV dose, given at Day 31 |  | 21

7. Secondary Outcome: Number of Participants With Solicited Systemic AEs After Each Vaccine Dose Administration
Description: The solicited systemic events after vaccination include fever (pyrexia), headache, fatigue, myalgia and arthralgia. Fever is defined as body temperature >=38 degree Celsius; preferred location for measuring the temperature is oral.
Time Frame: as for outcome 6
Population: Exposed set. Only those participants with solicited systemic AEs were included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Co-administration Group | Control Group
Number analyzed (Participants) | 538 | 546
Participants
  Fever, Dosing at Day 1 | 16 | 4
  Fever, Dosing at Day 31: number analyzed (Participants) | 0 | 510
  Fever, Dosing at Day 31 |  | 8
  Headache, Dosing at Day 1 | 144 | 83
  Headache, Dosing at Day 31: number analyzed (Participants) | 0 | 510
  Headache, Dosing at Day 31 |  | 97
  Fatigue, Dosing at Day 1 | 198 | 152
  Fatigue, Dosing at Day 31: number analyzed (Participants) | 0 | 510
  Fatigue, Dosing at Day 31 |  | 144
  Myalgia, Dosing at Day 1 | 176 | 89
  Myalgia, Dosing at Day 31: number analyzed (Participants) | 0 | 510
  Myalgia, Dosing at Day 31 |  | 108
  Arthralgia, Dosing at Day 1 | 80 | 41
  Arthralgia, Dosing at Day 31: number analyzed (Participants) | 0 | 510
  Arthralgia, Dosing at Day 31 |  | 67

8. Secondary Outcome: Number of Participants With Unsolicited AEs
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the administration of a study vaccine, which does not necessarily have a causal relationship with study vaccine. An unsolicited AE is an AE that is either not included in the list of solicited events or could be included in the list of solicited events but with an onset outside the specified period of follow-up for solicited events. Unsolicited AEs are communicated by participant/participant's caregiver(s) who have signed the informed consent. Unsolicited AEs include both serious adverse events (SAEs) and non-serious AEs.
Time Frame: Within 30 days (the day of vaccination and 29 subsequent days) after each vaccine administration (vaccines administered at Day 1 for Co-Administration Group and at Days 1 and 31 for Control group)
Population: Exposed set.
Measure: Count of Participants; unit: Participants
Arm/Group | Co-administration Group | Control Group
Number analyzed (Participants) | 553 | 557
Participants | 60 | 98

9. Secondary Outcome: Number of Participants With SAEs
Description: An SAE is defined as any untoward medical occurrence that results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is an important medical event.
Time Frame: Throughout the study period (from Day 1 up to 6 months after the last dose administration [last dose given at Day 1 for Co-administration Group and Day 31 for Control Group])
Population: Exposed set.
Measure: Count of Participants; unit: Participants
Arm/Group | Co-administration Group | Control Group
Number analyzed (Participants) | 553 | 557
Participants | 9 | 14

10. Secondary Outcome: Number of Participants With Potential Immune-mediated Diseases (pIMDs)
Description: The pIMD is a subset of AEs of special interest that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune etiology.
Time Frame: as for outcome 9
Population: Exposed set.
Measure: Count of Participants; unit: Participants
Arm/Group | Co-administration Group | Control Group
Number analyzed (Participants) | 553 | 557
Participants | 2 | 1

ADVERSE EVENTS:
Time Frame: Solicited AEs were collected up to Day 7 post each vaccination. Unsolicited AEs were collected up to Day 30 post each vaccination. SAEs and pIMDs were collected throughout the study period from Day 1 up to 6 months post last vaccination.
Description: Solicited and unsolicited events were reported per participant for the assessed timeframe (within 30 days after any vaccine dose administration) according to occurrence of each event, as pre-specified in Statistical Analysis Plan.
Arm/Group | Co-administration Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/553 | 2/557
Serious Adverse Events (participants affected / at risk) | 9/553 | 14/557
Other Adverse Events (participants affected / at risk) | 410/553 | 423/557
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Co-administration Group (N=553) | Control Group (N=557)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 2 (2)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2)
Necrotising fasciitis (Infections and infestations) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Fracture displacement (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Breast cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour rupture (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Co-administration Group (N=553) | Control Group (N=557)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiovascular disorder (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ear congestion (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Graves' disease (Endocrine disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Orbital haematoma (Eye disorders) | 1 (1) | 0 (0)
Swelling of eyelid (Eye disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 3 (3)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Periodontal inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
Axillary pain (General disorders) | 0 (0) | 1 (2)
Chills (General disorders) | 2 (3) | 1 (1)
Fatigue (General disorders) | 198 (245) | 217 (262)
Influenza like illness (General disorders) | 1 (1) | 1 (1)
Injection site erythema (General disorders) | 64 (85) | 48 (61)
Injection site pain (General disorders) | 337 (404) | 312 (365)
Injection site pruritus (General disorders) | 6 (6) | 2 (2)
Injection site swelling (General disorders) | 38 (49) | 38 (46)
Malaise (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 18 (20) | 13 (14)
Swelling (General disorders) | 0 (0) | 1 (2)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Acarodermatitis (Infections and infestations) | 0 (0) | 1 (1)
Arthritis infective (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2) | 3 (3)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1)
Coronavirus infection (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 11 (11)
Gastroenteritis (Infections and infestations) | 0 (0) | 4 (4)
Infective tenosynovitis (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 5 (5) | 4 (4)
Oral herpes (Infections and infestations) | 1 (1) | 4 (4)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 4 (4) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 7 (7)
Urinary tract infection (Infections and infestations) | 0 (0) | 5 (5)
Varicella zoster virus infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Soft tissue injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tooth dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fibrin D dimer increased (Investigations) | 1 (1) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 80 (100) | 94 (115)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 176 (205) | 157 (185)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 3 (3)
Dysgeusia (Nervous system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 144 (168) | 142 (175)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Sinus headache (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (3) | 0 (0)
Hypertonic bladder (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 2 (2)
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the full clinical trial.

DOCUMENTS (2):
  • Study Protocol (2023-06-23): https://cdn.clinicaltrials.gov/large-docs/07/NCT05879107/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-23): https://cdn.clinicaltrials.gov/large-docs/07/NCT05879107/SAP_001.pdf